CLINICAL TRIAL: NCT05588648
Title: A Phase I/II, Open-label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of Vactosertib as a Single Agent in Adolescents and Adults With Recurrent, Refractory or Progressive Osteosarcoma
Brief Title: Study to Assess Safety and Efficacy of Vactosertib in Adolescents and Adults With Recurrent, Refractory or Progressive Osteosarcoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedPacto, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-VAC-209
Record Dates: First submitted 2022-09-14; First posted 2022-10-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — vactosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): Single arm, open-label, no blinding or randomization procedure will be involved.
  Interventions: Drug: Vactosertib

INTERVENTIONS:
Drug: Vactosertib — Vactosertib is given twice a day, five days on and two days off in four-week cycles. Vactosertib is a transforming growth factor-beta (TGF-β) type 1 receptor inhibitor.
  Other Names: TEW-7197

SUMMARY:
MP-VAC-209 is a Phase I/II, open label, single arm, multi-center study to assess safety, tolerability, and antitumor activity of vactosertib as a single agent in adolescents and adults with recurrent, refractory, or progressive osteosarcoma. Vactosertib is given orally, twice a day, to people 12 years of age and older who meet the criteria for study enrollment.

DETAILED DESCRIPTION:
This is a Phase I/II, open label, single arm, proof of concept, multi-center (global) study to assess safety, tolerability, pharmacokinetics and antitumor activity of vactosertib as a Single Agent in Adolescents and Adults with Recurrent, Refractory or Progressive Osteosarcoma or bone lesions that have progressed, relapsed or are refractory to standard systemic therapy. Adolescents are defined as subjects aged 12 to <18-year-old.

During the Phase I part of the trial, dose limiting toxicity will be used to decide dose escalation according to the standard 3+3 rules to determine the maximum tolerated dose (MTD) and the recommended phase II dose (RP2D) in adults and adolescents.

Dose escalation will be conducted sequentially and independently in adults and adolescents, respectively. Dose escalation in adolescents will not start before dose escalation in adults is completed. Data from the Phase I part of the trail in adults will be reviewed by the DSMB before opening the Phase II part. Data from the Phase I in adolescents will be reviewed by the DSMB before each dose (de-)escalation. As soon as the RP2D in adolescents is established, adolescents will be enrolled in Phase II.

During Phase II, subjects will be enrolled at the RP2D determined independently for adults and adolescents. Data of the subjects enrolled in the Phase II will be pooled with data of subjects enrolled at the same dose level during Phase I to evaluate the efficacy in a total of 42 adult and adolescent subjects.

In all parts of the study, the DSMB will convene upon occurrence of a grade 5 or any two sequentially occurring grade 4 drug related adverse events. In such case, accrual may not resume unless the DSMB has conducted a review and offered a recommendation to continue the study.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all the following inclusion criteria to be eligible for enrollment:

Informed Consent/Assent Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Age ≥12 years at the time of screening

Type of Subject and Disease Characteristics

1. Subjects may be male or female and must be equal to or greater than 12 years of age. No large studies have evaluated the use of vactosertib in younger pediatric subjects, for this reason, children younger than 12 years of age are excluded from this study.
2. Subjects must have histologic verification of Osteosarcoma (OS)
3. Subjects must have measurable disease per RECIST 1.1 (Appendix C), documented by clinical, radiographic and histologic criteria, and have progressed, relapsed or become refractory to conventional therapy.
4. Subjects must have recovered from the acute toxic effects with ≤ Grade 1 as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0 of all prior chemotherapy and immunotherapy with the exception of alopecia, anorexia, bone pain, and tumor pain prior to entering this study.
5. Myelosuppressive chemotherapy: Must have adequate recovery of counts from previous treatment prior to entry onto this study.
6. Inclusion criteria include adequate renal function, ECOG performance status 0-2, and either Lansky performance status of 50-100% (<16 years old), or Karnofsky performance status 50-100% (≥16 years old). Subjects who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
7. Subjects must have normal organ and marrow function as defined below:

   a. Adequate bone marrow function defined as: i. Peripheral absolute neutrophil count (ANC) ≥ 750/mcL ii. Platelet count ≥ 75,000/mcL (transfusion independent) iii. Hemoglobin ≥ 8.0 g/dL (may receive packed red blood cell transfusions) b. Adequate liver function defined as: i. Total bilirubin ≤ 1.5 times the upper limit of normal for age ii. AST (SGOT) and ALT (SGPT) 2.5 X institutional upper limit of normal iii. Albumin (serum or plasma) > 2 g/dL c. Adequate cardiac function defined as: i. Ejection fraction of ≥ 50% by echocardiogram or MUGA
8. Subjects must have the ability to understand and the willingness to sign a written informed consent document if ≥ 18 years of age and an assent document if < 18 years of age (per country).
9. Renal laboratory inclusion:
10. Relapsed osteosarcoma (first, second, third or any relapse, subject who have recovered from chemotherapy and any other investigational drug/agent treatment, radiotherapy or surgical procedure), with histological confirmed diagnosis of osteosarcoma at original presentation, and progressive disease documented by imaging within 3 months of entry into the trial.

Exclusion Criteria

The subject must be excluded from participating in the trial if:

1. Subjects who have moderate or severe cardiovascular disease

   1. Subjects who have uncontrolled intercurrent illness, including but not limited to, ongoing or active infection requiring systemic therapy, symptomatic congestive heart failure (New York Heart Association Class III/IV), uncontrolled hypertension (≥150/90mmHg), unstable angina pectoris or myocardial infarction (≤ 6 months prior to screening), uncontrolled cardiac arrhythmia, clinically significant cardiac valvulopathy requiring treatment, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the subject to give written informed consent
   2. Subjects who have major abnormalities at the Investigator's discretion based on electrocardiogram (ECG)and Doppler ECHO and MUGA results at screening or within 14 days before screening. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms in both male and female calculated from 12-lead ECGs.
   3. Subjects who have increase in brain natriuretic peptide (BNP) or increase in troponin (over 99th percentile upper reference limit) at Screening (based on the normal range of relevant study center)
   4. Subjects who have risk factors for ascending aortic aneurysm such as genetic disorder and trauma and risk factors for aortic stenosis
   5. Subjects who have a history of heart or aorta surgery
2. Subjects who have clinically significant gastrointestinal bleeding within 4 weeks before screening
3. Subjects who have a known history or suspected hypersensitivity to any excipients of the investigational product.
4. Subjects who have received prior treatment targeting the signaling pathway of TGF-β
5. Subjects who have a disease or condition that affects the mechanism of the investigational product, or are currently using or planning to use:

   1. Drugs that are exclusively or primarily eliminated by cytochrome P-450 isozyme (CYP) including CYP1A2, CYP2D6, CYP2B6, or CYP3A4 (Concurrent use of drugs that are known potent CYP3A4 inducers including but not limited to Phenytoin, Rifampin, and St. John's wort. Concurrent use of foods that are known strong CYP3A4 inhibitors including but not limited to grapefruit juice, Itraconazole, Ketoconazole, Lopinavir/ritonavir, Mibefradil, and Voriconazole. The topical use of these medications (if applicable), such as 2% ketoconazole cream, may be allowed.)
   2. Drugs that are exclusively or primarily eliminated by UDP glucuronyltransferase (UGT) 1A1 (UGT1A1)
   3. Drugs that are substrates for the drug transporter multidrug resistance protein 1 (MDR1) have a narrow therapeutic window or are strong inhibitors of drug transporter MDR1
6. Subjects who are unable to swallow tablets
7. Subjects who have a history of or are suspected of drug abuse
8. Female subjects of child-bearing potential who have a positive result on a pregnancy test at screening or are unable to agree to use an effective barrier method of birth control to avoid pregnancy during the study period (e.g., sterilization, intrauterine contraceptive device, combination of oral contraception and barrier contraception, combination of other hormone delivery systems and barrier contraception, contraceptive cream, combination of cream, jelly, or form and diaphragm or condom). Male subjects of reproductive potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 90 days after the last dose of study therapy.
9. Subjects, in the opinion of the Investigator, who are unsuitable to participate in the study
10. Subjects who were treated with other investigational products within 28 days before screening or within a period shorter than 5-times the half-life of the investigational product
11. Subjects currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study drug Note: Subjects who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
12. Subjects taking prohibited medications when using vactosertib as following. A minimal washout period of 5 half-lives for the following drugs is recommended prior to the first dosing
13. Subjects with a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. HIV-positive subjects and HIV-positive subjects on antiretroviral therapy are ineligible because of the risk for developing a lethal infection when treated with immunosuppressive therapy.
15. Concurrent active/acute infection.
16. Non-metastatic osteosarcoma (OS) for whom standard therapy are possible at the time of the study may be excluded.
17. Chronic use of corticosteroids or other immunosuppressive agents. Note: High dose is defined as a prescription of >5 mg oral prednisolone and long term as duration of treatment >1 month (based on NICE. Corticosteroids - oral (accessed Apr 2017).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dose finding associated with the overall nature and severity of AEs associated with treatment. | Assessment of adverse events and laboratory abnormalities. through study completion, an average of 1 year
  Maximum tolerated dose (MTD) and recommended dose (RD)

SECONDARY OUTCOMES:
Overall survival. | Acquiring the measures associated with phase I/phase II primary endpoints.
  Overall survival (1 year) calculated from date of enrollment to the dates of documented evidence of progression or death up to 12 months.
Time to response(TTR) | Post two cycle of treatment, evaluation. through study completion, an average of 1 year.
  To evaluate the time to response(TTR) from Vactosertib treatment to show PR or CR. To characterize the pharmacokinetics(PK) of Vactosertib to 6 patients assigned to dose- escalation phase and the firsts 12 patients assigned to the dose expansion phase.

CONTACTS AND LOCATIONS:
Locations (3):
- UH Rainbow Babies & Children's Hospital, Cleveland, Ohio, United States
- South Korea (2):
  - National Cancer Center, Gyeonggi-do
  - Korea Institute of Radiological & Medical Sciences, Seoul

IPD SHARING:
Plan to Share IPD: No